CLINICAL TRIAL: NCT07297745
Title: Trial of Aldosterone-hybrid SteRoid for Guiding curablE Treatment of Primary Aldosteronism (TARGET-PA)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: Singapore General Hospital (Other); Sengkang General Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TARGET-PA
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Hyperaldosteronism; Primary; Primary Aldosteronism Due to Aldosterone Producing Adenoma
Keywords: Hybrid hormone; Subtyping; adrenalectomy; adrenal vein sampling; biomarkers; steroid profiling
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Intervention Model Description: The investigators will prospectively recruit participants with primary aldosteronism who are keen for surgery if unilateral disease is diagnosed. Participants will undergo both routine subtyping (adrenal vein sampling and/or molecular imaging) and research subtyping (blood tests for hybrid hormone coupled with computed tomography). All results will be reviewed at a multi-disciplinary meeting, with computed tomography discussed first (radiologist will be masked to results of hybrid hormones and adrenal vein sampling), then hybrid hormones, then adrenal vein sampling. Participants with either adrenal vein sampling lateralization, or elevated hybrid hormones with a unilateral adrenal nodule and normal contralateral gland on computed tomography will be offered surgery. All participants will be re-evaluated post-surgery for biochemical cure of primary aldosteronism (co-primary outcome). Genetic sequencing will be performed on resected adrenals for KCNJ5 mutation (co-primary outcome).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid hormones (Experimental): Previous studies have shown that hybrid hormones are elevated in patients with unilateral primary aldosteronism who have large, visible adenomas in their adrenal glands. These tumors harbour a somatic KCNJ5 mutation and are also most likely to be cured of hypertension after surgery.
  Hence, the investigators hypothesize that high hybrid hormones levels, in the presence of an adenoma on a computed tomography imaging would identify study participants who can proceed to surgery.
  Interventions: Diagnostic Test: Hybrid hormones

INTERVENTIONS:
Diagnostic Test: Hybrid hormones — Participants will have a baseline blood sample taken so the investigators can measure the adrenal steroid biomarkers 18-oxocortisol, 18-hydroxylcortisol and other steroids.
  The collected plasma or serum will then be analyzed in the laboratory using validated methods, such as liquid chromatography-tandem mass spectrometry (LC-MS/MS), to determine the levels of these biomarkers.

SUMMARY:
The goal of this project is to improve the diagnostic pathway for patients with primary aldosteronism, by validating non-invasive biomarkers coupled with routine computed tomography imaging. The aim is to reduce reliance on invasive procedures, shorten diagnostic timelines, and enhance accessibility to definitive diagnosis and treatment globally.

DETAILED DESCRIPTION:
Primary Aldosteronism is a common but under-diagnosed condition, despite being a curable cause of secondary hypertension with significant long-term health consequences if left untreated. Once the diagnosis of primary aldosteronism is confirmed, subtype tests are required to demonstrate unilateral primary aldosteronism before curative surgery. Most patients need to undergo adrenal vein sampling, an invasive procedure performed under radiological guidance. However, this procedure is technically-challenging, with failure to cannulate both adrenal veins frequently leading to inconclusive results. Many patients worldwide may be offered surgery based on computed tomography imaging alone because of a lack of adrenal vein sampling expertise or a failed adrenal vein sampling result.

High hybrid hormones indicate a functional KCNJ5-mutant aldosterone-producing adenoma and, when coupled with computed tomography imaging, may provide a non-invasive alternative to adrenal vein sampling for identifying unilateral primary aldosteronism.

Ultimately, this trial aims to reduce the number of patients that will require an invasive adrenal vein sampling in future clinical diagnostics. This will improve access, and allow more patients to receive timely and curative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary aldosteronism according to the Endocrine Society guideline 2025.
* Willing to undergo subtype testing with adrenal vein sampling and/or molecular imaging (Positron Emission Tomography/Computed Tomography, PET/CT).
* Keen for surgical treatment if shown to have unilateral primary aldosteronism.

Exclusion Criteria:

* Inability to provide written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with complete biochemical success after unilateral adrenalectomy for unilateral primary aldosteronism using Primary Aldosteronism Surgical Outcome (PASO) measured at least six months post-adrenalectomy. | 6 months
  Proportion of participants with correction of hypokalaemia and normalisation of aldosterone-renin-ratio following unilateral adrenalectomy, as per PASO criteria.
Proportion of participants with KCNJ5-mutant aldosterone producing adenoma/nodule | 6 months
  Proportion of participants with histopathology and genetic confirmation of KCNJ5-mutant aldosterone producing adenoma/nodule in resected adrenals.

SECONDARY OUTCOMES:
Proportion of participants with complete clinical success after unilateral adrenalectomy for unilateral primary aldosteronism using Primary Aldosteronism Surgical Outcome (PASO) measured at least six months post-adrenalectomy. | 6 months
  Proportion of participants with reduction in blood pressure and reduction anti-hypertensive medication following unilateral adrenalectomy, as per PASO criteria.
Cost-effectiveness of using hybrid hormones coupled with computed tomography imaging versus other subtyping tests including adrenal vein sampling and/or molecular imaging in diagnosing participants with unilateral primary aldosteronism | 6 months
  Cost-effectiveness of the diagnostic course will be calculated by using calculated costs per quality-adjusted life years (QALYs)
Diagnostic criteria using hybrid hormones/ steroid profiling coupled with computed tomography imaging | 6 months
  The criteria of hybrid hormones/ steroid profiling coupled with computed tomography imaging which offer the best sensitivity and specificity for lateralization of aldosterone-producing adenoma.

CONTACTS AND LOCATIONS:
Overall Officials: Troy Puar, FRCP, PhD, Principal Investigator — Changi General Hospital
Locations (4):
- Singapore (4):
  - Changi General Hospital, Singapore, Singapore
  - National University Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Singapore General Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No